CLINICAL TRIAL: NCT04267328
Title: Post-Operative Cognitive Dysfunction in Normal Aging Patients Undergoing Elective Orthopedic Surgery
Acronym: POCD
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A19-224
Record Dates: First submitted 2020-02-11; First posted 2020-02-12 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having surgery: Older adults undergoing elective orthopedic surgery.
  Interventions: Procedure: Elective Orthopedic Surgery

INTERVENTIONS:
Procedure: Elective Orthopedic Surgery — Patients having knee (unilateral primary osteoarthritis or bilateral primary osteoarthritis) surgery, hip (unilateral primary osteoarthritis or bilateral primary osteoarthritis) or shoulder (primary osteoarthritis) elective surgery.

SUMMARY:
Post-operative cognitive dysfunction (POCD) is a common concern for aging patients undergoing elective orthopedic surgery and significantly effects health outcomes. This study aims to evaluate the incidence of and risk factors associated with post-operative cognitive dysfunction in aging patients without prior history for mild cognitive impairment or dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 and ≤90
* Any patient undergoing elective orthopedic surgery for hip, knee, or shoulder replacement (as defined by diagnostic codes: M16.0, M16.12, M16.11, M17.0, M17.12, M17.11, M19.011, M19.012)

Exclusion Criteria:

* History of cognitive impairment of dementia
* Montreal cognitive assessment (MoCA) <26
* History of Parkinson's disease, progressive supranuclear palsy, corticobasal degeneration, normal pressure hydrocephalus, Huntington's disease, stroke, seizure disorder, brain tumor, or brain surgery
* History of surgery requiring anesthesia within the past 3 months

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Regions Hospital orthopedics center in Saint Paul, MN with a scheduled surgery fitting the diagnostic codes listed in the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Having Surgery
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Having Surgery
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Presence of Post Operative Cognitive Dysfunction (POCD)
Description: Defined as a decline of 1.5 or greater standard deviation on any one of the cognitive test performed from baseline to three-months post surgery. Score range: 0-100. A higher score indicates more cases of incident of POCD.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Having Surgery
Number analyzed (Participants) | 47
Participants | 15

ADVERSE EVENTS:
Time Frame: 3 months from end of surgery
Arm/Group | Patients Having Surgery
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04267328/Prot_SAP_000.pdf